CLINICAL TRIAL: NCT01049971
Title: Reduction of Wound Infections in Laparoscopic Colon Resections by Wound Protectors
Brief Title: REDWIL: Reduction of Wound Infections in Laparoscopic Colon Resections by Wound Protectors
Acronym: REDWIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: PD Dr. JP Ritz, Dr. JC Lauscher, Charité Campus Benjamin Franklin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA4/089/07
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2007-12

CONDITIONS: Colorectal Surgery; Wound Infections
Keywords: colorectal surgery; wound infection; wound protector; laparoscopy; surgical site infection after laparoscopic colorectal surgery with minilaparotomy
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- no wound protector (Active Comparator): instead of wound protector, a woven drape is applied
  Interventions: Device: no wound protector
- wound protector (Experimental): after minilaparotomy, wound protector is applied
  Interventions: Device: wound protector

INTERVENTIONS:
Device: wound protector — after minilaparotomy, the wound protector is applied
  Other Names: Vi-Drape (Trademark) wound protector
  Arms: wound protector
Device: no wound protector — use of woven drape instead of wound protector
  Arms: no wound protector

SUMMARY:
Surgical site infection is common in colorectal surgery leading to increased postoperative pain, longer hospital stay, delayed wound healing and increased re-operation rates. Hence, reducing the wound infection rate is a major aim in abdominal surgery.

Wound protectors were invented for retracting the abdominal wall and keeping the abdominal wall sterile in order to reduce bacterial colonialization of the wound and wound infections.

This is a prospective-randomized trial comparing use of wound protectors versus woven drapes in laparoscopic colon resections with minilaparotomy.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic colorectal resection with minilaparotomy

Exclusion Criteria:

* emergency operation
* patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2007-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
percentage of wound infections | 6 months postoperatively
  the total percentage of wound infections within 6 months postoperatively will be analyzed

SECONDARY OUTCOMES:
colonialization of abdominal wall with bacteria | 6 months postoperatively
  a swab of the abdominal wall is taken before skin closure routinely in every participating patient and the bacteria found is analyzed
postoperative costs | 6 months postoperatively
  the costs for the operation, for the hospital stay including re-admissions, and for the outpatient stay is analyzed
length of hospital stay | 6 months postoperatively
  the total hospital stay including re-admissions is analyzed
cosmetic result | 6 months postoperatively
  the satisfaction with the cosmeti result is analyzed in every patient by questionnaire 6 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Campus Benjamin Franklin; Hindenburgdamm 30, Berlin, State of Berlin, Germany